CLINICAL TRIAL: NCT07106528
Title: Organoid-Based Drug Sensitivity Model Guided Personalized Precision Treatment for Extensive-Stage Small Cell Lung Cancer: A Prospective, Multicenter, Randomized Controlled Trial
Brief Title: Organoid-guided vs Topotecan Therapy in Relapsed Extensive-Stage Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K8538
Record Dates: First submitted 2025-07-22; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Extensive-stage Small Cell Lung Cancer (ES-SCLC); Extensive-stage Small Cell Lung Cancer (SCLC); Small Cell Lung Cancer ( SCLC )
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Topotecan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Organoid-Guided Personalized Therapy (Experimental): Drug selection based on organoid drug sensitivity testing
  Interventions: Drug: Organoid Drug Sensitivity Testing-Guided Therapy
- Standard Topotecan Chemotherapy (Active Comparator): Intravenous topotecan
  Interventions: Drug: Topotecan

INTERVENTIONS:
Drug: Organoid Drug Sensitivity Testing-Guided Therapy — Personalized drug selection (chemotherapy/targeted therapy/immunotherapy) based on ex vivo organoid drug response testing
  Arms: Organoid-Guided Personalized Therapy
Drug: Topotecan — Intravenous topotecan 1.25 mg/m² daily on days 1-5 of each 21-day cycle
  Arms: Standard Topotecan Chemotherapy

SUMMARY:
This study aims to provide personalized treatment options for patients with extensive-stage small cell lung cancer (SCLC) whose disease has worsened after initial chemotherapy.

Researchers will use a novel approach called "tumor organoid drug sensitivity testing":

A small sample of the patient's tumor (from biopsy or fluid) is grown into miniature 3D tumor models ("organoids") in the lab.

These organoids are exposed to various FDA-approved second-line drugs (including chemotherapy and newer targeted/immunotherapy drugs if available).

The most effective drug for each patient's organoids will be recommended for their treatment.

128 participants will be randomly assigned to one of two groups:Experimental Group: Receive organoid-guided personalized therapy; Control Group: Receive standard second-line chemotherapy (Topotecan).

The study will compare: How long the cancer remains controlled (Progression-Free Survival); Overall survival time; Treatment response rates and side effects.

Potential benefits: May identify more effective treatments for individual patients; Could extend time without cancer progression.

Risks: Organoid testing requires an additional tumor biopsy/fluid collection; Possible side effects from second-line drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older.
2. Pathologically confirmed extensive-stage small cell lung cancer (ES-SCLC) (AJCC 9th edition, Stage IV).
3. Previously received first-line platinum-based systemic chemotherapy and experienced recurrence or progression during first-line treatment or within ≤ 6 months after completion of first-line treatment.
4. Availability of sufficient tumor tissue or malignant serous effusion for organoid culture.
5. Presence of measurable lesions based on RECIST 1.1.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
7. Adequate bone marrow and organ function, confirmed by baseline blood count, blood biochemistry, and urine biochemistry tests.
8. Asymptomatic and stable central nervous system (CNS) metastases are allowed.
9. Expected survival of at least 3 months.
10. For male participants: Agreement to use effective contraception during treatment and for at least 180 days after the last dose of study treatment; prohibition of sperm donation during this period.
11. For female participants: Not pregnant or breastfeeding, and meeting at least one of the following:

    Women of non-childbearing potential; or Agreement to use effective contraception during treatment and for at least 180 days after the last dose of study treatment; or Women of childbearing potential must have a negative serum or urine pregnancy test (with a minimum sensitivity of 25 IU/L or HCG equivalent units) within 72 hours before initiating treatment.
12. Voluntary participation with signed informed consent and willingness to comply with study follow-up procedures.

Exclusion Criteria:

1. Mixed tumor pathology or lack of histological confirmation.
2. Previous receipt of second-line or higher systemic anti-tumor therapy for ES-SCLC.
3. Symptomatic or progressive brain metastases, or meningeal metastases.
4. History of other malignant tumors that are progressive or require active treatment within the past 5 years.
5. Presence of active infections, severe organ dysfunction, or other contraindications to anti-tumor treatment.
6. Inability to obtain tumor tissue or insufficient malignant serous effusion for collection.
7. Expected survival of less than 3 months.
8. Inability to complete standardized clinical diagnosis/treatment or regular follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From date of randomization until the date of first documented progression (RECIST v1.1) or death from any cause, whichever occurs first, assessed up to 100 months.
  From the date of randomization to the date of first recording of disease progression ( RECIST v1.1 ) or all-cause death, whichever occurred first.

SECONDARY OUTCOMES:
Overall Survival (OS) | From date of randomization until the date of death from any cause, assessed up to 100 months.
  From date of randomization until the date of death from any cause
Objective Response Rate (ORR) | From date of randomization until the date of first documented progression, assessed by RECIST v1.1 criteria at 6- to 8-week intervals up to 100 months.
  From date of randomization until the date of first documented progression, assessed by RECIST v1.1 criteria at 6- to 8-week
Duration of Response (DOR) | From date of first documented objective response (CR or PR per RECIST v1.1) until the date of first documented progression or death from any cause, whichever occurs first, assessed up to 100 months.
  From date of first documented objective response (CR or PR per RECIST v1.1) until the date of first documented progression or death from any cause, whichever occurs first
Grade ≥3 Adverse Events | From date of first treatment administration until 3 months after last dose, assessed by CTCAE v5.0 criteria.
  The incidence of treatment-related adverse events ≥ grade 3 ( CTCAE v5.0 ).